CLINICAL TRIAL: NCT01634347
Title: Memory Reconsolidation Blockade for Treating Drug Addiction: a Feasibility Study
Brief Title: Memory Reconsolidation Blockade for Treating Drug Addiction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Alain Brunet, Ph.D., Sponsor-Investigator, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRPL-004
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Substance Dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol and memory reactivation (Experimental)
  Interventions: Drug: Propranolol and memory reactivation
- Placebo and memory reactivation (Placebo Comparator)
  Interventions: Drug: Placebo and memory reactivation

INTERVENTIONS:
Drug: Propranolol and memory reactivation — Propranolol will be administered once a week for a 3 or 6 week period. Each propranolol administration will be followed by memory reactivation.
  Arms: Propranolol and memory reactivation
Drug: Placebo and memory reactivation — Placebo will be administered once a week for a 3 or 6 week period. Each placebo administration will be followed by memory reactivation.
  Arms: Placebo and memory reactivation

SUMMARY:
The treatment involves administering propranolol, a medication indicated for treating high blood pressure. Propranolol is hypothesized to reduce the strength of drug or alcohol cravings (an integral factor involved in relapse), specifically when memories of substance use are recalled. In this study, propranolol or a placebo will be administered to patients participating in a drug or alcohol rehabilitation facility once a week over three or six weeks. After receiving propranolol or placebo, strong memories associated with substance craving are recalled by asking participants to read aloud a summary of a substance use experience. The investigators hypothesize that participants who receive propranolol will report fewer and less intense drug or alcohol cravings than participants who receive the placebo or treatment-as-usual.

DETAILED DESCRIPTION:
Trial Objectives: To test the feasibility of reconsolidation blockade as an adjunct treatment for reducing drug or alcohol cravings in individuals diagnosed with a substance dependence or substance abuse disorder and participating in a drug rehabilitation program.

Study Design and Duration: This study will be a 3 to 6 week, randomized, double-blind trial involving participants with a DSM-IV-TR diagnosis of substance dependence or abuse. Consented participants meeting enrolment criteria will receive a dose of propranolol (1mg/kg) or placebo ninety minutes before undergoing a brief memory reactivation procedure twice a week for a three-week period (or once a week for a six week period, depending on the participants availability) as an adjunct to their usual drug rehabilitation treatment. Participants will be randomized to one of two treatment arms (i.e. placebo group + treatment as usual, or propranolol group + treatment as usual) and remain in that arm for the duration of the study. Participants from the placebo arm will be offered the opportunity to continue receive open-label propranolol treatment for another 3-6 weeks following the double-blind phase of the study. A four-month follow-up assessment will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age
* Female subjects must not be of child bearing potential or be non pregnant and be established on an acceptable method of birth control or be one who abstains from sex
* Diagnosis of substance dependence or substance abuse disorder within a 1-month period prior to screening
* Currently enrolled in a drug rehabilitation treatment program for marijuana, cocaine, heroin, other opiates, benzodiazepine, alcohol, or amphetamine addictions
* Individuals who consent to remain abstinent from all drugs of abuse (except nicotine) and from alcohol for 24 hours prior to enrolment and for the duration of the study
* Individuals treated with the following medications must be on stable doses for at least 1-month prior to the screening visit and during the entire study: anxiolytics, sedatives, hypnotics, antidepressants, antipsychotics
* Individuals taking Selective Serotonin Reuptake Inhibitors (SSRIs) or Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs) must accept to skip their morning dose the day of each study visit
* Individuals shall not start taking new medications on a regular basis during the study
* Fluency in French or English

Exclusion Criteria:

* Systolic blood pressure <100 mm Hg
* Cardiac rhythm below 55 beats per minute
* A medical condition that contraindicates the administration of propranolol
* Previous adverse reaction to, or non-compliance with, beta-blocker
* Current use of medication that may involve potentially dangerous interactions with propranolol.
* Women who are pregnant or breast feeding
* Past or present bipolar disorder or psychosis
* Individuals with current dependence on any substance besides, cocaine, heroin, other opiates, benzodiazepines, amphetamines, marijuana, or alcohol
* Subjects judged as being at significant risk of self injurious/suicidal or violent/homicidal behavior
* Participation in another drug trial within 30 days prior to the screening visit or during the study
* Any condition that can significantly affect the absorption of the study medication
* Presence of any clinical condition that might interfere with the interpretation of the efficacy and safety results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Substance craving scales | Weeks 3 or 6
  The craving scales ask about current craving for substances. Items for the questionnaires represent distinct conceptualizations of substance craving: (1) desire to use; (2) anticipation of positive outcomes from use; (3) anticipation of relief from withdrawal symptoms or relief from negative mood; (4) intention and planning to use; (5) lack of control over use.

SECONDARY OUTCOMES:
Number of days in a drug or alcohol addiction rehabilitation treatment program | Once or twice a week for a 3-to-6 week period, as well as at 4 months post-baseline
Addiction severity | Once or twice a week for a 3-to-6 week period, as well as at 4 months post-baseline
Rates of successfully completing a drug or alcohol rehabilitation program | Once or twice a week for a 3-to-6 week period, as well as at 4 months post-baseline
Rates of planned or unplanned departure and expulsion from a drug or alcohol rehabilitation program | Once or twice a week for a 3-to-6 week period, as well as at 4 months post-baseline
Frequency and intensity of drug or alcohol cravings | Once or twice a week for a 3-to-6 week period
Brief psychiatric rating scale | Once or twice a week for a 3-to-6 week period, as well as at 4 months post-baseline
Rates of relapse of drug or alcohol dependence a drug or alcohol rehabilitation program. | Once or twice a week for a 3-to-6 week period, as well as at 4 months post-baseline
Rates of adverse events | From baseline to 28 days after the last administration of study medication

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Heritage Home Drug and Alcohol Rehabilitation Centre, Godmanchester, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec

REFERENCES:
- See also: Related Info — http://www.sobriety.ca